CLINICAL TRIAL: NCT02758561
Title: 2015 Motivational Interviewing in Women's Pelvic Wellness Education Project
Brief Title: Motivational Interviewing in Women's Pelvic Wellness Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20150564-01H
Record Dates: First submitted 2015-12-22; First posted 2016-05-02 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Pelvic Floor Disorders; Urinary Incontinence (UI); Pelvic Prolapse Conditions
Keywords: decisional aid; workshops; urinary incontinence; pelvic organ prolapse; pelvic floor dysfunction; decisional conflict
MeSH Terms: conditions — Pelvic Floor Disorders; Urinary Incontinence; Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (No Intervention): Standard of care
- Workshop (Experimental): 90 minute workshop on either Urinary Incontinence (UI) or Pelvic Organ Prolapse (POP)
  Interventions: Behavioral: Workshop

INTERVENTIONS:
Behavioral: Workshop — The first 15 minutes will be an information session on either Urinary Incontinence (UI) or Pelvic Organ Prolapse (PO) led by a Nurse Continence Advisor.
  The following 60 minutes will comprise a psychologist-led group discussion. The structured discussion will encourage participants to share experiences, thoughts, and feelings on pelvic floor disorders. Resistances and barriers to seeking treatment will be discussed. Decision-making processes will be explored.
  During the final 15 minutes, participants will be asked to complete a survey to evaluate the workshop. The survey will assess satisfaction with the information provided, quality of group discussion, comfort level with the group experience, and their satisfaction with the roles of the nurse continence advisor and psychologist.
  Arms: Workshop

SUMMARY:
This pilot study will assess the feasibility and acceptability of an educational workshop on pelvic floor disorders and its potential impact on decisional conflict.

DETAILED DESCRIPTION:
Pelvic floor disorders can significantly affect a woman's quality of life, yet many feel uncomfortable openly discussing these topics. Treatments include lifestyle modification, medications, and/or surgery. "Decisional conflict" arises when patients have difficulty choosing between several viable treatment options. Factors contributing to decisional conflict include biased information, poor peer support, and unaddressed fears. Effective counselling may help address these factors.

There are few studies on how decision coaching can help women with prolapse and incontinence reach a satisfactory decision about treatment. This study aims to use the principals of shared decision making to address decisional conflict surrounding treatment for pelvic floor disorders. Specifically, the investigators will evaluate the feasibility and acceptability of small group workshops on pelvic organ prolapse and urinary incontinence led by a nurse continence advisor and a psychologist (decision coach).

Results of this study will inform future development of interdisciplinary, patient-centered approaches to enhanced decision making in women's health.

ELIGIBILITY:
Inclusion Criteria:

* Women ages >18 years old
* Urinary incontinence and/or pelvic organ prolapse
* First visit with urogynecologist

Exclusion Criteria:

* Anal incontinence
* Previous pelvic radiation therapy
* Requirement for a Substitute Decision Maker
* Inability to attend the workshop
* Unwilling to attend an English-language workshop
* Unwilling to complete English-language surveys

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05; Primary Completion 2017-05 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Change in "Decisional Conflict" between baseline and followup, as measured by the Decisional Conflict Scale (O'Connor 1995). | The Decisional Conflict Scale (DCS), will be administered to participants in the control and intervention groups at baseline and first follow up visit, approx. 3 months later.
  The decisional conflict scale (DCS) is a validated scale that measures (a) perceived uncertainty between options, (b) factors contributing to uncertainty (feeling uninformed, unclear about values, unsupported in decision making), and (c) factors contributing to effective decision making (feeling the choice is informed, values-based, likely to be implemented, and satisfaction with the decision). 13 A total decisional conflict score from 0 (no decisional conflict) to 100 (extremely high decisional conflict) is given, as well as five sub-scores for each factor listed above.

SECONDARY OUTCOMES:
Participant satisfaction with the workshop. | This will be measured using a survey administered to participants immediately following the workshop
  Non-validated questionnaire addressing participants' perceived satisfaction with the following aspects of the workshop: group discussion, the information session, and the workshop as a whole. In addition there are four free text questions: 1) What changes will you make in your decision for treatment as a result of this workshop?; 2)Tell us about one thing you found most valuable in this workshop; 3)What would you change about this workshop?; 4) Other comments

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Schachter, MD, FRCSC, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Riverside Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT02758561/Prot_SAP_000.pdf